CLINICAL TRIAL: NCT01262638
Title: A Placebo-Controlled, Randomized, Double-Blind, Parallel Group, Multicenter Study to Evaluate the Efficacy and Safety of ETC-1002 in Subjects With Hypercholesterolemia and Either Normal or Elevated Triglycerides.
Brief Title: A Study to Assess the Efficacy and Safety of ETC-1002 in Subjects With Elevated Blood Cholesterol and Either Normal or Elevated Triglycerides
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Esperion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ETC-1002-003
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Results first posted 2021-03-16 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- ETC-1002 120 mg (Group 1) (Experimental): Subjects with hypercholesterolemia and normal triglycerides
  Interventions: Drug: ETC-1002
- ETC-1002 80 mg (Group 2) (Experimental): Subjects with hypercholesterolemia and normal triglycerides
  Interventions: Drug: ETC-1002
- ETC-1002 40 mg (Group 3) (Experimental): Subjects with hypercholesterolemia and normal triglycerides
  Interventions: Drug: ETC-1002
- Placebo (Group 4) (Experimental): Subjects with hypercholesterolemia and normal triglycerides
  Interventions: Drug: Placebo
- ETC-1002 120 mg (Group 5) (Experimental): Subjects with hypercholesterolemia and elevated triglycerides
  Interventions: Drug: ETC-1002
- ETC-1002 80 mg (Group 6) (Experimental): Subjects with hypercholesterolemia and elevated triglycerides
  Interventions: Drug: ETC-1002
- ETC-1002 40 mg (Group 7) (Experimental): Subjects with hypercholesterolemia and elevated triglycerides
  Interventions: Drug: ETC-1002
- Placebo (Group 8) (Experimental): Subjects with hypercholesterolemia and elevated triglycerides
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ETC-1002 — ETC-1002 daily for 12 weeks
  Arms: ETC-1002 120 mg (Group 1); ETC-1002 120 mg (Group 5); ETC-1002 40 mg (Group 3); ETC-1002 40 mg (Group 7); ETC-1002 80 mg (Group 2); ETC-1002 80 mg (Group 6)
Drug: Placebo — Placebo daily for 12 weeks
  Arms: Placebo (Group 4); Placebo (Group 8)

SUMMARY:
This Phase 2 proof-of-concept study will assess the lipid regulating efficacy and safety of ETC-1002 in subjects with hypercholesterolemia and either normal or elevated triglycerides.

ELIGIBILITY:
Major Inclusion Criteria:

* Provision of written informed consent prior to any study-specific procedure
* Fasting LDL-C between 130 and 220 mg/dL following wash-out of all lipid regulating medications and supplements
* Fasting triglyceride <400 mg/dL following wash-out of all lipid regulating medications and supplements
* BMI between 18 and 35 mg/kg2

Major Exclusion Criteria:

* Clinically significant cardiovascular disease, diabetes or uncontrolled hypertension
* Females of child bearing potential (i.e., females who are not surgically sterile or post-menopausal)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2010-12; Primary Completion 2011-08-23 (Actual); Study Completion 2011-08-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Chandler, Arizona
  - Greenbrae, California
  - Santa Rosa, California
  - Jacksonville, Florida
  - Chicago, Illinois
  - Iowa City, Iowa
  - Louisville, Kentucky
  - Kalamazoo, Michigan
  - Raleigh, North Carolina
  - Houston, Texas
  - Richmond, Virginia

REFERENCES:
- [Result] Ballantyne CM, Davidson MH, Macdougall DE, Bays HE, Dicarlo LA, Rosenberg NL, Margulies J, Newton RS. Efficacy and safety of a novel dual modulator of adenosine triphosphate-citrate lyase and adenosine monophosphate-activated protein kinase in patients with hypercholesterolemia: results of a multicenter, randomized, double-blind, placebo-controlled, parallel-group trial. J Am Coll Cardiol. 2013 Sep 24;62(13):1154-62. doi: 10.1016/j.jacc.2013.05.050. Epub 2013 Jun 13. PMID 23770179

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 177 participants were enrolled and treated across 11 study sites in the United States.
Pre-assignment Details: During Screening, appropriate participants washed off all lipid-regulating drugs and supplements as necessary for 6 weeks prior to randomization. Participants not taking lipid-regulating medications or supplements for 4 weeks prior to Screening may have combined the S1 and Q1 visits. Participants with hypercholesterolemia were stratified into the normal (<150 milligrams per deciliter [mg/dL]) or elevated (≥150 mg/dL) triglycerides (TG) stratum.
Groups:
- ETC-1002 40 mg: Participants received ETC-1002 40 milligrams (mg), orally, once daily for 12 weeks.
- ETC-1002 80 mg: Participants received ETC-1002 80 mg, orally, once daily for 12 weeks.
- ETC-1002 120 mg: Participants received ETC-1002 120 mg, orally, once daily for 12 weeks.
- Placebo: Participants received placebo, orally, once daily for 12 weeks.
Period: Overall Study
Arm/Group | ETC-1002 40 mg | ETC-1002 80 mg | ETC-1002 120 mg | Placebo
Started | 45 | 44 | 44 | 44
Completed | 38 | 38 | 38 | 37
Not Completed | 7 | 6 | 6 | 7
Not completed — Adverse Event | 3 | 4 | 3 | 4
Not completed — Protocol Violation | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 1
Not completed — Per Investigator/Sponsor/Regulatory Body | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 1
Not completed — Participant Went Out of Town | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data are reported for members of the Safety Population, comprised of all randomized participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | ETC-1002 40 mg | ETC-1002 80 mg | ETC-1002 120 mg | Placebo | Total
Number analyzed (Participants) | 45 | 44 | 44 | 44 | 177
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.4 (8.66) | 58.8 (9.00) | 56.7 (9.92) | 55.5 (10.40) | 57.3 (9.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 21 | 19 | 13 | 79
  Male | 19 | 23 | 25 | 31 | 98
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1 | 2
  Black or African American | 7 | 7 | 2 | 6 | 22
  White | 38 | 36 | 41 | 37 | 152
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Calculated Low-density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] — Baseline was defined as the mean of the values from Weeks -1 and 0.
  milligrams per deciliter (mg/dL) | 163.1 (24.88) | 170.2 (26.23) | 165.0 (23.08) | 167.4 (22.03) | 166.4 (24.05)
LDL-C by Triglyceride (TG) Stratum [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the mean of the values from Weeks -1 and 0. Population: The Overall Number of Baseline Participants analyzed is the sum of the participants in the Normal Stratum and Elevated Stratum.
  mg/dL
    Normal Stratum, TG<150 mg/dL: number analyzed (Participants) | 23 | 22 | 22 | 22 | 89
    Normal Stratum, TG<150 mg/dL | 153.8 (22.06) | 164.6 (25.36) | 160.2 (17.30) | 166.6 (17.87) | 161.2 (21.15)
    Elevated Stratum, TG≥150 mg/dL: number analyzed (Participants) | 22 | 22 | 22 | 22 | 88
    Elevated Stratum, TG≥150 mg/dL | 172.9 (24.35) | 175.7 (26.46) | 169.8 (27.25) | 168.2 (25.94) | 171.7 (25.73)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 12 in Calculated Low-Density Lipoprotein-Cholesterol (LDL-C)
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline was defined as the mean of the values from Weeks -1 and 0. Least square (LS) mean percent change from Baseline to Week 12 was based on an analysis of covariance (ANCOVA) model with effects of treatment and triglyceride (TG) stratum and Baseline value as a covariate. Missing LDL-C values at Week 12 were imputed using the last observation carried forward (LOCF) procedure (only post-Baseline values were carried forward).
Time Frame: Baseline; 12 weeks
Population: Modified Intent-to-Treat (mITT) Population: all randomized participants who received at least 1 dose of study medication and had a Baseline assessment and at least 1 post-Baseline assessment, excluding any assessments taken more than 2 days after a dose of study medication
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 40 mg | ETC-1002 80 mg | ETC-1002 120 mg | Placebo
Number analyzed (Participants) | 42 | 44 | 42 | 42
Percent Change | -17.9 (2.17) | -25.0 (2.12) | -26.6 (2.16) | -2.1 (2.16)
Statistical Analysis 1: Comparison: ETC-1002 40 mg vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Difference in Least Squares Means = -15.7, 95% CI 2-sided [-21.8 to -9.7]
Statistical Analysis 2: Comparison: ETC-1002 80 mg vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Difference in Least Squares Means = -22.9, 95% CI 2-sided [-28.9 to -16.9]
Statistical Analysis 3: Comparison: ETC-1002 120 mg vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Difference in Least Squares Means = -24.5, 95% CI 2-sided [-30.5 to -18.4]

2. Primary Outcome: Percent Change From Baseline to Week 12 in LDL-C by Triglyceride (TG) Stratum
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline was defined as the mean of the values from Weeks -1 and 0. LS mean percent change from Baseline to Week 12 was based on an ANCOVA model with effects of treatment and center and Baseline value as a covariate. Missing LDL-C values at Week 12 were imputed using the LOCF procedure (only post-Baseline values were carried forward).
Time Frame: Baseline; 12 weeks
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Groups:
- ETC-1002 40 mg: Participants received ETC-1002 40 mg, orally, once daily for 12 weeks.
Arm/Group | ETC-1002 40 mg | ETC-1002 80 mg | ETC-1002 120 mg | Placebo
Number analyzed (Participants) | 42 | 44 | 42 | 42
Percent Change
  Normal (TG<150 mg/dL): number analyzed (Participants) | 20 | 22 | 22 | 20
  Normal (TG<150 mg/dL) | -17.8 (2.92) | -21.9 (2.73) | -29.2 (2.72) | 0.3 (2.89)
  Elevated (TG≥150 mg/dL): number analyzed (Participants) | 22 | 22 | 20 | 22
  Elevated (TG≥150 mg/dL) | -17.8 (3.21) | -28.1 (3.22) | -23.6 (3.37) | -4.5 (3.22)

3. Secondary Outcome: Percent Change From Baseline to Week 12 in TG
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline was defined as the mean of the values from Weeks -1 and 0. LS mean percent change from Baseline to Week 12 was based on an ANCOVA model with effects of treatment and TG stratum and Baseline value as a covariate. Missing TG values at Week 12 were imputed using the LOCF procedure (only post-Baseline values were carried forward).
Time Frame: Baseline; 12 weeks
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 40 mg | ETC-1002 80 mg | ETC-1002 120 mg | Placebo
Number analyzed (Participants) | 42 | 44 | 42 | 42
Percent Change | -15.1 (4.29) | -10.6 (4.16) | 1.1 (4.26) | -1.2 (4.29)

4. Secondary Outcome: Percent Change From Baseline to Week 12 in High-Density Lipoprotein-Cholesterol (HDL-C)
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline was defined as the mean of the values from Weeks -1 and 0. LS mean percent change from Baseline to Week 12 was based on an ANCOVA model with effects of treatment and TG stratum and Baseline value as a covariate. Missing HDL-C values at Week 12 were imputed using the LOCF procedure (only post-Baseline values were carried forward).
Time Frame: Baseline; 12 weeks
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 40 mg | ETC-1002 80 mg | ETC-1002 120 mg | Placebo
Number analyzed (Participants) | 42 | 44 | 42 | 42
Percent Change | 7.2 (2.22) | 0.9 (2.12) | 4.4 (2.16) | 2.4 (2.18)

5. Secondary Outcome: Percent Change From Baseline to Week 12 in Non-HDL-C
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline was defined as the mean of the values from Weeks -1 and 0. LS mean percent change from Baseline to Week 12 was based on an ANCOVA model with effects of treatment and TG stratum and Baseline value as a covariate. Missing non-HDL-C values at Week 12 were imputed using the LOCF procedure (only post-Baseline values were carried forward).
Time Frame: Baseline; 12 weeks
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 40 mg | ETC-1002 80 mg | ETC-1002 120 mg | Placebo
Number analyzed (Participants) | 42 | 44 | 42 | 42
Percent Change | -17.4 (2.01) | -22.7 (1.95) | -23.0 (2.00) | -2.3 (2.00)

6. Secondary Outcome: Percent Change From Baseline to Week 12 in Total Cholesterol (TC)
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline was defined as the mean of the values from Weeks -1 and 0. LS mean percent change from Baseline to Week 12 based on an ANCOVA model with effects of treatment and TG stratum and Baseline value as a covariate. Missing TC values at Week 12 were imputed using the LOCF procedure (only post-Baseline values were carried forward).
Time Frame: Baseline; 12 weeks
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 40 mg | ETC-1002 80 mg | ETC-1002 120 mg | Placebo
Number analyzed (Participants) | 42 | 44 | 42 | 42
Percent Change | -11.5 (1.53) | -17.8 (1.50) | -17.1 (1.53) | -1.4 (1.53)

7. Secondary Outcome: Percent Change From Baseline to Week 12 in Apolipoprotein B (ApoB)
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline was defined as the value from Week 0. LS mean percent change from Baseline to Week 12 was based on an ANCOVA model with effects of treatment and TG stratum and Baseline value as a covariate. Missing ApoB values at Week 12 were imputed using the LOCF procedure (only post-Baseline values were carried forward).
Time Frame: Baseline; 12 weeks
Population: mITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 40 mg | ETC-1002 80 mg | ETC-1002 120 mg | Placebo
Number analyzed (Participants) | 39 | 39 | 38 | 39
Percent Change | -14.6 (1.83) | -18.4 (1.82) | -22.1 (1.84) | -0.9 (1.83)

8. Secondary Outcome: Percent Change From Baseline to Week 12 in Apolipoprotein AI (ApoAI)
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline was defined as the mean of the values from Week 0. LS mean percent change from Baseline to Week 12 was based on an ANCOVA model with effects of treatment and TG stratum and Baseline value as a covariate. Missing ApoAI values at Week 12 were imputed using the LOCF procedure (only post-Baseline values were carried forward).
Time Frame: Baseline; 12 weeks
Population: mITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 40 mg | ETC-1002 80 mg | ETC-1002 120 mg | Placebo
Number analyzed (Participants) | 39 | 39 | 38 | 39
Percent Change | 2.9 (1.96) | -2.7 (1.95) | 0.0 (1.97) | -3.1 (1.95)

9. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipoprotein (a)
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline was defined as the mean of the values from Week 0. LS mean percent change from Baseline to Week 12 was based on an ANCOVA model with effects of treatment and TG stratum and Baseline value as a covariate. Missing Lipoprotein (a) values at Week 12 were imputed using the LOCF procedure (only post-Baseline values were carried forward).
Time Frame: Baseline; 12 weeks
Population: mITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 40 mg | ETC-1002 80 mg | ETC-1002 120 mg | Placebo
Number analyzed (Participants) | 39 | 39 | 38 | 39
Percent Change | 0.3 (5.20) | 7.6 (5.20) | 16.2 (5.27) | -2.7 (5.22)

10. Secondary Outcome: Percent Change From Baseline to Week 12 in Free Fatty Acids (FFA)
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline was defined as the mean of the values from Week 0. LS mean percent change from Baseline to Week 12 was based on an ANCOVA model with effects of treatment and TG stratum and Baseline value as a covariate. Missing FFA values at Week 12 were imputed using the LOCF procedure (only post-Baseline values were carried forward).
Time Frame: Baseline; 12 weeks
Population: mITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 40 mg | ETC-1002 80 mg | ETC-1002 120 mg | Placebo
Number analyzed (Participants) | 39 | 40 | 37 | 40
Percent Change | 2.5 (6.15) | -14.4 (6.08) | 5.3 (6.34) | 3.6 (6.09)

11. Secondary Outcome: Percent Change From Baseline to Week 12 in High-Sensitivity C-Reactive Protein (hsCRP)
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline was defined as the mean of the value from Week 0. LS mean percent change from Baseline to Week 12 was based on an ANCOVA model with effects of treatment and TG stratum and Baseline value as a covariate. Missing hsCRP values at Week 12 were imputed using the LOCF procedure (only post-Baseline values were carried forward).
Time Frame: Baseline; 12 weeks
Population: mITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 40 mg | ETC-1002 80 mg | ETC-1002 120 mg | Placebo
Number analyzed (Participants) | 39 | 39 | 38 | 39
Percent Change | 18.4 (42.45) | 57.0 (42.44) | 48.0 (43.24) | 86.6 (42.45)

12. Secondary Outcome: Percent Change From Baseline to Week 12 in Total LDL Particles
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline was defined as the mean of the values from Week 0. LS mean percent change from Baseline to Week 12 was based on an ANCOVA model with effects of treatment and TG stratum and Baseline value as a covariate. Missing values at Week 12 were imputed using the LOCF procedure (only post-Baseline values were carried forward).
Time Frame: Baseline; 12 weeks
Population: mITT Population. Only participants with available date were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 40 mg | ETC-1002 80 mg | ETC-1002 120 mg | Placebo
Number analyzed (Participants) | 39 | 40 | 36 | 40
Percent Change | -14.8 (2.26) | -16.3 (2.23) | -20.7 (2.34) | 1.9 (2.22)

13. Secondary Outcome: Percent Change From Baseline to Week 12 in Total HDL Particles
Description: as for outcome 12
Time Frame: Baseline; 12 weeks
Population: mITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 40 mg | ETC-1002 80 mg | ETC-1002 120 mg | Placebo
Number analyzed (Participants) | 39 | 40 | 36 | 40
Percent Change | 5.7 (1.78) | 3.6 (1.74) | 7.3 (1.84) | 0.4 (1.75)

14. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were defined as adverse events (AEs) that began or worsened in severity after the first dose of study medication, occurring up to 30 days after the last dose of study medication.
Time Frame: up to 12 weeks
Population: Safety Population: all randomized participants who received at least 1 dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | ETC-1002 40 mg | ETC-1002 80 mg | ETC-1002 120 mg | Placebo
Number analyzed (Participants) | 45 | 44 | 44 | 44
Participants | 34 | 32 | 31 | 33

15. Secondary Outcome: Number of Participants With Clinically Significant Physical Examination Findings
Description: Clinical significance was determined by the investigator.
Time Frame: up to 12 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | ETC-1002 40 mg | ETC-1002 80 mg | ETC-1002 120 mg | Placebo
Number analyzed (Participants) | 45 | 44 | 44 | 44
Participants | 2 | 2 | 0 | 2

16. Secondary Outcome: Number of Participants With Clinically Important Changes From Baseline in Vital Sign Values
Description: Clinical importance was determined by the investigator.
Time Frame: Baseline; up to 12 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | ETC-1002 40 mg | ETC-1002 80 mg | ETC-1002 120 mg | Placebo
Number analyzed (Participants) | 45 | 44 | 44 | 44
Participants | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Clinically Important Changes From Baseline in Electrocardiogram Values
Description: Clinical importance was determined by the investigator.
Time Frame: Baseline; up to 12 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | ETC-1002 40 mg | ETC-1002 80 mg | ETC-1002 120 mg | Placebo
Number analyzed (Participants) | 45 | 44 | 44 | 44
Participants | 0 | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With the Indicated Abnormal Laboratory Parameter Values at Week 12
Description: Laboratory abnormalities are laboratory values that are outside the normal range.
Time Frame: Week 12
Population: Safety Population. Only participants with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | ETC-1002 40 mg | ETC-1002 80 mg | ETC-1002 120 mg | Placebo
Number analyzed (Participants) | 45 | 44 | 44 | 44
Participants
  Alanine aminotransferase: number analyzed (Participants) | 38 | 39 | 39 | 37
  Alanine aminotransferase | 4 | 3 | 3 | 4
  Aspartate aminotransferase: number analyzed (Participants) | 38 | 39 | 39 | 37
  Aspartate aminotransferase | 5 | 6 | 8 | 2
  Creatine kinase: number analyzed (Participants) | 38 | 39 | 39 | 37
  Creatine kinase | 12 | 8 | 3 | 5
  Creatinine: number analyzed (Participants) | 38 | 39 | 39 | 37
  Creatinine | 1 | 0 | 1 | 0
  Total bilirubin: number analyzed (Participants) | 38 | 39 | 39 | 37
  Total bilirubin | 1 | 1 | 0 | 1
  Uric acid: number analyzed (Participants) | 38 | 39 | 39 | 37
  Uric acid | 6 | 8 | 6 | 3
  Hemoglobin: number analyzed (Participants) | 39 | 39 | 38 | 37
  Hemoglobin | 5 | 8 | 4 | 2
  Leukocytes: number analyzed (Participants) | 39 | 39 | 38 | 37
  Leukocytes | 3 | 2 | 1 | 1

ADVERSE EVENTS:
Time Frame: up to 12 weeks
Description: Treatment-emergent adverse events (TEAEs), defined as adverse events (AEs) that began or worsened in severity after the first dose of study medication, occurring up to 30 days after the last dose of study medication, are reported. The analysis was performed using the Safety Population, comprised of all randomized participants who received at least 1 dose of study medication.
Arm/Group | ETC-1002 40 mg | ETC-1002 80 mg | ETC-1002 120 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/44 | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/44 | 0/44 | 1/44
Other Adverse Events (participants affected / at risk) | 15/45 | 18/44 | 17/44 | 17/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ETC-1002 40 mg (N=45) | ETC-1002 80 mg (N=44) | ETC-1002 120 mg (N=44) | Placebo (N=44)
Chest Pain (General disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ETC-1002 40 mg (N=45) | ETC-1002 80 mg (N=44) | ETC-1002 120 mg (N=44) | Placebo (N=44)
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 1 | 3
Nausea (Gastrointestinal disorders) | 3 | 3 | 4 | 2
Fatigue (General disorders) | 3 | 1 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 3 | 1 | 1
Urinary Tract Infection (Infections and infestations) | 4 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 1
Headache (Nervous system disorders) | 5 | 5 | 7 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No